CLINICAL TRIAL: NCT03816098
Title: The Accuracy of Chinese Version of Swallowing Disturbance Questionnaire in Screening Inpatient Elderly
Brief Title: The Accuracy of Swallowing Disturbance Questionnaire in Screening Inpatient Elderly
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Hsiao-chan, Lai, Speech-language therapist, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Other Study IDs: 07-XD-080
Record Dates: First submitted 2019-01-21; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Deglutition Disorders
Keywords: elderly; screening
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- elderly patients with dysphagia
- elderly patients without dysphagia

SUMMARY:
The aim of this research was to examine the accuracy of translated Chinese version of Swallowing Dysphagia Questionnaire and to evaluate the prevalence of dysphagia and its clinical manifestation in patients over 65 years old.

ELIGIBILITY:
Inclusion Criteria:

* (1) age over 65 years old; (2) does not use enteral tube feeding; (3) no serious mental or cognitive conditions; no aphasia

Exclusion Criteria:

* (1) age under 65; (2) use enteral tube feeding; (3) subjects with serious mental or cognitive conditions or aphasia (4) Allergy to barium sulfate suspension

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 40 elderly inpatients age over 65 are included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-02-11 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Swallowing Disturbance Questionnaire | At the baseline
  Chinese version of Swallowing Dysphagia Questionnaire consists of 15 questions regarding oral and pharyngeal stage of dysphagia. Subjects are asked to fill out the questionnaire concerning current state and during the past year using a 4-point scale.
Videofluroscopy Swallowing Study (VFSS) | At the baseline
  VFSS studies are conducted using 4 different consistencies: thin liquid, nectar-thick liquid, puree, and cookie. Subjects are asked to take 2 trials for each consistency to assess if any oral or pharyngeal dysphagia occurs.

SECONDARY OUTCOMES:
Clinical water test | At the baseline
  Each subject takes 3 trials of 3cc-water using a dropper. Then sequential water drinking is assessed (about 60-70 ml). We assess: coughing, choking, voice changes. At least one symptom means dysphagia.
Mini-Mental State Examination (MMSE) | At the baseline
  Mini-Mental State Examination was used to identify subjects' cognitive state.The following four cut-off levels should be employed to classify the severity of cognitive impairment: no cognitive impairment=24-30; mild cognitive impairment=19-23; moderate cognitive impairment=10-18; and severe cognitive impairment<9.